CLINICAL TRIAL: NCT05184036
Title: Development of an ICT Platform-Awareness System for the Support of Low Vision
Acronym: LIFE4LV
Status: Active, not recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Vasileios Karampatakis, Professor, Aristotle University Of Thessaloniki
Other Study IDs: T1EDK-03742
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Low Vision Digital Assistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Low Vision — * The application of a questionnaire evaluating the functionality and quality of life and records several of the daily life of Greek LV patients.
  * The evaluation of the basic parameters of visual function included in the LIFE4LV platform in order to evaluate the effectiveness of this platform in correlation with the routine ophthalmologic exams.
  * The evaluation of existing digital supportive tools for LV and record of the patient's feedback

SUMMARY:
Low Vision (LV) has a detrimental impact on Quality of Life (QoL) of affected individual's and is considered a major healthcare problem according to World Health Organization. The primary objective of this study is the development of an integrated ICT platform-awareness system for the assistance of individuals with LV for the evaluation of visual ability. It is of high importance to develop and apply appropriate strategies aiming at the improvement of daily living and access to healthcare services of patients with LV. Secondary objectives are the evaluation of a suite of supportive mobile applications (magnification, reading, etc)'' for individuals with LV in order to improve their ability to perform daily activities and the development of a new questionnaire to assess the functionality and quality of life of individuals with LV.Investigators will conduct an effectiveness study to determine if the features of LIFE4LV platform provide low vision patients and their physicians with appropriate benefits.

DETAILED DESCRIPTION:
Low Vision (LV) refers to a significant impairment of vision without the possibility of improvement by any therapeutic intervention, affecting significantly the abilities of LV individuals. In the 10th revision of the WHO International Statistical Classification of Diseases, Injuries and Causes of Death, 'low vision' is defined as visual acuity of less than 6/18 but equal to or better than 3/60, or a corresponding visual field loss to less than 20°, in the better eye with the best possible correction.

The aim of the current study is to explore innovative strategies to support individuals with LV using new digital technologies developed in the field of information and these applications to assist these patients.

The development of a patient digital file is an additional part of innovation since the possible changes during the course of the disease could be detected and recorded.

Specifically, the current study aims at the development of an integrated ICT platform-awareness system for the support of LV individuals, including a digital platform for the evaluation of visual ability of LV patients in concert with their physician.

Specifically, objectives of the study are:

* The development of the digital platform consisted of applications assessing basic parameters of the visual function. The platform aims to improve the level of patient's follow up and communication with their physician and does not replace the physical examination in any case.
* Additionally, the election of supportive mobile applications (magnification, reading, etc)'' for individuals with LV in a form of a supportive suite of digital tools may facilitate the performance of basic activities.
* Another objective is the design and validation of a new questionnaire to assess the functionality and the quality of life of Greek individuals with LV.
* The development of a training handbook/manual is also considered as an important parameter to provide patients with appropriate instructions for the correct use of the assistive digital tools and applications. The above manual aims to improve the utilization of the digital platform and the suite, as some parameters should be evaluated under the appropriate conditions and requires a period of education, especially when individuals are not familiar with digital media

ELIGIBILITY:
Inclusion Criteria

1. Visual acuity in the better-seeing eye 20/50-20/400
2. Visual field at least 10 degrees
3. Informed written consent to the processing of personal data

Exclusion Criteria:

1. Younger than 18 years of age
2. Severe mental disorder (any type of dementia, under medication that affects mental function, etc.) or neurological problems that cause difficulty in communication
3. End-stage diseases (chronic kidney disease, cancer, liver failure, etc.), which may affect their performance and their ability
4. Severe mobility problems
5. Active or rapidly progressive eye disease in an acute phase that can affect directly visual performance e.g. intravitreal hemorrhage
6. Ocular diseases causing reversible visual impairment (e.g. cataract, uncorrected refractive errors etc.)
7. Not receiving topical or systemic treatment with known toxic effects on the lens, retina or optic nerve (e.g. ethambutol, chloroquine or hydroxychloroquine, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with LV according to WHO definition (10th edition, WHO International Statistical Classification of Diseases, Injuries and Causes of Death)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Design of a digital platform for the evaluation of basic parameters of visual function | Baseline
  The efficacy of a new digital color test will be evaluated in terms of its validity properties in identifying acquired color vision defects. Other basic parameters of the visual ability will also be included in the digital, LIFE4LV platform and be evaluated for their efficacy to serve as a useful tool both for LV patients and their physicians.
The evaluation of the usability of a set of supportive digital applications | Baseline
  The evaluation of the usability of supportive digital applications (magnification, text reading etc)
  The expected outcomes would be:
  * Feedback from participants regarding the usability of supportive applications for LV
  * Better communication and interaction between LV individuals and their physician
  * Relief and less burden on their familiars
  * Better level of independence
  * Enhanced opportunity to engage in social and other activities
  * Improvement of their mental state to the extent that this can be achieved
Design and Validation of the LIFE4LV questionnaire for the Greek population | Baseline
  A new questionnaire will be developed and evaluated for its phychometric properties for the assessment of the functionality and QoL of LV patients in Greece

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Karampatakis, Prof., Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Central Macedonia, Greece

REFERENCES:
- [Result] Karampatakis V, Almaliotis D, Talimtzi P, Almpanidou S. Design and Validation of a Novel Smartphone-Based Visual Acuity Test: The K-VA Test. Ophthalmol Ther. 2023 Jun;12(3):1657-1670. doi: 10.1007/s40123-023-00697-x. Epub 2023 Mar 24. PMID 36961662
- [Result] Gkioka M, Almpanidou S, Lioti N, Almaliotis D, Karampatakis V. Daily Functionality of People with Low Vision: The Impact of Visual Acuity, Depression, and Life Orientation-A Cross-Sectional Study. Behav Neurol. 2024 Feb 26;2024:4366572. doi: 10.1155/2024/4366572. eCollection 2024. PMID 38440066
- [Result] Karampatakis V, Almaliotis D, Papadopoulou EP, Almpanidou S. Design of a novel smartphone-based photostress recovery time test for detecting abnormalities in the macula. A cross-sectional study. Ann Med Surg (Lond). 2022 Apr 29;77:103699. doi: 10.1016/j.amsu.2022.103699. eCollection 2022 May. PMID 35638075
- [Result] Almaliotis D, Almpanidou S, Chatzimbalis T, Nikolaidou A, Talimtzi P, Karampatakis V. Correlation between color vision, visual acuity, contrast sensitivity and photostress recovery in the visually impaired: a cross-sectional study. Ann Med Surg (Lond). 2023 Nov 20;86(2):742-747. doi: 10.1097/MS9.0000000000001522. eCollection 2024 Feb. PMID 38333302
- [Result] Almpanidou S, Almaliotis D, Karamitopoulos L, Topouzis F, Konstas AG, Labiris G, Dardavesis T, Fountoulakis KN, Chatzisavvas KC, Karampatakis V. Development and Validation of the Life for Low Vision Questionnaire (LIFE4LVQ) Using Rasch Analysis: A Questionnaire Evaluating Ability and Independence. J Clin Med. 2023 Mar 28;12(7):2549. doi: 10.3390/jcm12072549. PMID 37048633
- [Result] Karampatakis V, P Papadopoulou E, Almpanidou S, Karamitopoulos L, Almaliotis D. Evaluation of contrast sensitivity in visually impaired individuals using K-CS test. A novel smartphone-based contrast sensitivity test-Design and validation. PLoS One. 2024 Feb 8;19(2):e0288512. doi: 10.1371/journal.pone.0288512. eCollection 2024. PMID 38330096
- [Result] Karampatakis V, Almaliotis D, Karamitopoulos L, Kalliris G, Almpanidou S. A Novel Smartphone-Based Color Test for Detection of Color Vision Defects in Age Related Macular Degeneration. J Ophthalmol. 2022 Mar 31;2022:9744065. doi: 10.1155/2022/9744065. eCollection 2022. PMID 35399161